CLINICAL TRIAL: NCT02768740
Title: Double Blinded, Randomized Trial, Comparing Intravenous Bolus of 50 mg of Hydrocortisone Every 6 Hours for 7 Days With a Continuous Infusion of 300 mg Per Day of Hydrocortisone 300-mg Group During 5 Days in the Treatment of Septic Shock.
Brief Title: Hydrocortisone 50 mg Every 6 Hours Compared to Hydrocortisone 300 mg Per Day in Treatment of Septic Shock.
Acronym: HSHC00582434
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association Niçoise de Réanimation Médicale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-005824-34
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — hydrocortisone hemisuccinate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 200 mg group (Active Comparator): Patients received an intravenous bolus of 50 mg of hydrocortisone every six hours for seven days associated with a continuous infusion of placebo for five days.
  Interventions: Drug: Hydrocortisone hemisuccinate
- 300 mg group (Experimental): Patients received an initial bolus of 100 mg of hydrocortisone followed by a continuous infusion of 300 mg per day for five days associated with a bolus of placebo every six hours for seven days.
  Interventions: Drug: Hydrocortisone hemisuccinate

INTERVENTIONS:
Drug: Hydrocortisone hemisuccinate — In the 200-mg group, patients received an intravenous bolus of 50 mg of hydrocortisone every six hours for seven days associated with a continuous infusion of placebo for five days. In the 300-mg group, patients received an initial bolus of 100 mg of hydrocortisone followed by a continuous infusion of 300 mg per day for five days associated with a bolus of placebo every six hours for seven days.
  Other Names: Saline solution as placebo

SUMMARY:
We performed a multicenter, prospective, randomized, double-blind, pilot study in four adult medical intensive care units. Patients presenting septic shock were rapidly administered one of two regimens of hydrocortisone, either a 50-mg intravenous bolus every six hours during seven days (200-mg group) or a 100-mg initial bolus followed by a continuous infusion of 300 mg daily for five days (300-mg group). Hydrocortisone was stopped abruptly at the end of treatment.

DETAILED DESCRIPTION:
Hydrocortisone hemisuccinate (Hydrocortisone Upjohn) was supplied as a powder in 100 mg vials to be reconstituted with 2 ml of sterile water diluent. The placebo was saline serum supplied as 10 ml ampoules. The study drugs were administered according to two protocols. In the 200-mg group, patients received an intravenous bolus of 50 mg of hydrocortisone every six hours for seven days associated with a continuous infusion of placebo for five days. In the 300-mg group, patients received an initial bolus of 100 mg of hydrocortisone followed by a continuous infusion of 300 mg per day for five days associated with a bolus of placebo every six hours for seven days. In the two groups, hydrocortisone was stopped abruptly at the end of treatment. The investigators had the choice or resuming hydrocortisone at the end of the fifth day if deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* septic shock in accordance with the American College of Chest Physicians/Society of Critical Care Medicine Consensus Committee criteria. Septic shock was managed in accordance with the 2004 edition of the Surviving Sepsis Campaign guidelines.
* no minimal vasopressor dose was needed to enter the trial.

Exclusion Criteria:

* medical history of adrenal insufficiency
* ongoing corticosteroid treatment
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mortality | 28-day
  The primary end point was to determine a difference in 28-day mortality between the 200-mg and 300-mg groups.

SECONDARY OUTCOMES:
Incidence of permanent shock between groups | 28-day
  Permanent shock (PS) was defined as permanent catecholamine support (epinephrine or norepinephrine) in the ICU, from the onset of septic shock to death without a period of reversal.
Incidence of shock relapse between groups | 28-day
  Shock relapse (SR) was defined as recurrence of septic shock requiring catecholamine resumption.
Incidence of post hydrocortisone hemodynamic rebound between groups | 28-day
  Post hydrocortisone hemodynamic rebound (PHHR) was defined as SR within 48 hours after hydrocortisone cessation.
Incidence of adverse events between groups. | 28-day
  Incidences of hemorrhagic events, superinfections and the amount of needed insulin were compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Bernardin, M.D., Principal Investigator — Association Niçoise de Réanimation Médicale

IPD SHARING:
Plan to Share IPD: Undecided
The data are available for additional analysis